CLINICAL TRIAL: NCT02089360
Title: Study of Serum Level of Advanced Glycated Endproducts and Development of Coronary Atherosclerosis in Patients Undergoing Coronary Angiogram
Brief Title: Adavanced Glycated Endproducts and Development of CAD
Acronym: AGENDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhang Qi, MD, Director, Cardiac Catheterization Lab, Shanghai Jiao Tong University School of Medicine
Other Study IDs: RJH20140311
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Atherosclerosis; Inflammation
Keywords: Advanced glycation end product; coronary; atherosclerosis; inflammation; outcome
MeSH Terms: conditions — Atherosclerosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood sample is taken for all patients underwent coronary angiogram after getting informed consent, and stored in requested condition, for measuring serum levels of different kinds of factors.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Blood sample is prospectively taken from consecutive patients underwent coronary angiogram in our center, after getting informed consent from the patients. Serum level of advanced glycation end products (AGEs) was measured and the clinical features of patients (including angiographic results) were entered into our database. Clinical follow-up was performed for all patients, and the relationship between AGEs and paitents' outcome were analyzed. Further intervention will be adjusted according to the results,including clinical and basic research in lab.

DETAILED DESCRIPTION:
Serum levels of HMGB1, HMGB2, ADAM10, etc. will be measured in lab and animal studies will be designed to intervene the adverse interaction between abnormal serum concentration of AGEs, etc. and worse clinical results.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent coronary angiogram for suspected coronary artery disease and potential percutaneous coronary intervention

Exclusion Criteria:

* patients underwent coronary angiogram for other reasons, including pre-surgery examination
* patients with severe co-morbidity, and life expectancy less than one-year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent coronary angiogram
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 5-year
  including death, occurrence of myocardial infarction, and coronary revascularization

SECONDARY OUTCOMES:
progression in coronary atherosclerosis | 5-year
  repeated coronary angiogram in patients with symptom aggravation or occurrence of myocardial infarction, to evaluate the progression of coronary lesions, comparing to the baseline results.

OTHER OUTCOMES:
Serum level of AGEs | baseline
  serum levels of AGEs will be measured and the relationship between clinical outcomes will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yang CD, Shen Y, Lu L, Yang ZK, Hu J, Zhang RY, Shen WF, Ding FH, Wang XQ. Visit-to-visit HbA1c variability is associated with in-stent restenosis in patients with type 2 diabetes after percutaneous coronary intervention. Cardiovasc Diabetol. 2020 Sep 4;19(1):133. doi: 10.1186/s12933-020-01111-7. PMID 32887588
- [Derived] Yang CD, Shen Y, Ding FH, Yang ZK, Hu J, Shen WF, Zhang RY, Lu L, Wang XQ. Visit-to-visit fasting plasma glucose variability is associated with left ventricular adverse remodeling in diabetic patients with STEMI. Cardiovasc Diabetol. 2020 Sep 2;19(1):131. doi: 10.1186/s12933-020-01112-6. PMID 32878604
- [Derived] Yang CD, Shen Y, Lu L, Ding FH, Yang ZK, Zhang RY, Shen WF, Jin W, Wang XQ. Insulin resistance and dysglycemia are associated with left ventricular remodeling after myocardial infarction in non-diabetic patients. Cardiovasc Diabetol. 2019 Aug 7;18(1):100. doi: 10.1186/s12933-019-0904-3. PMID 31391045